CLINICAL TRIAL: NCT06452082
Title: Retrospective Observational Study on the Risk in Developing Long-COVID Syndrome After Acute COVID-19 Disease and in Contracting SARS-CoV-2 Infection After COVID-19 Vaccination in Relation to Vitamin D3 Supplementation in Outpatients of Endocrinology Department
Brief Title: Retrospective Observational Study on the Risk in Developing Long-COVID Syndrome and in Contracting SARS-CoV-2 Infection After COVID-19 Vaccination in Relation to Vitamin D3 Supplementation
Acronym: LONGVITAVAX2
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Di Filippo, Medical Physician Specialist in Endocrinology, IRCCS San Raffaele
Other Study IDs: ABIO/NC/06
Record Dates: First submitted 2024-06-06; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Vitamin d Deficiency; COVID-19; Long COVID
MeSH Terms: conditions — Vitamin D Deficiency; COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients on therapy with cholecalciferol
- patients not on cholecalciferol therapy

SUMMARY:
The aim of this observational retrospective study is to evaluate the effect of supplementation with cholecalciferol D3 in reducing the risk of:

* occurence of Long COVID syndrome after acute COVID-19 illness
* occurence of SARS-CoV-2 infection after anti-COVID-19 vaccination

DETAILED DESCRIPTION:
Anamnestic, laboratory and therapeutic data will be collected during outpatient visits.

ELIGIBILITY:
Inclusion Criteria (For aim I):

* age ≥18
* outpatient with first visit on Endocrinology Department performed from 01/01/2020 to 31/12/2022
* previous SARS CoV-2 infection
* clinical,anamnestic and therapeutic data 6 months post SARS CoV-2 infection
* data on cholecalciferol supplementation
* signature of informed consent

Exclusion Criteria (For aim I):

* age ≤ 18
* pregnant or breastfeeding women
* patients suffering from primary and/or acquired immunodeficiency and/or severe impairment of general clinical conditions
* patients treated with drugs that interfere with vitamin D metabolism
* first vaccination anti Sars COVID performed before the acute infection
* first vaccination performed within 6 months of the acute infection
* patients unable to sign the informed consent

Inclusion Criteria (For aim 2)

-- age ≥18

* outpatient with first visit on Endocrinology Department performed from 01/01/2020 to 31/12/2022
* vaccination with BNT162b2 Biontec mRNA Pfizer/BioNtech
* clinical, anamnestic and therapeutic data 6 months post SARS CoV-2 infection
* data on cholecalciferol supplementation
* signature of informed consent

Exclusion Criteria (For aim 2):

* age ≤ 18
* pregnant or breastfeeding women
* patients suffering from primary and/or acquired immunodeficiency and/or severe impairment of general clinical conditions
* patients treated with drugs that interfere with vitamin D metabolism
* additional vaccination performed before 6-12 months
* acute infection before the vaccination
* patients unable to sign the informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: outpatients affected by endocrine-metabolic disease with first visit to the Endocrinology Unit carried out between 01/01/2020 and 12/31/2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Analyse the rates of Long COVID syndrome occurance after acute COVID-19 disease in patients treated with and without cholecalciferol. | to 01/01/2020 from 31/12/2022
  Analyse the rates of Long COVID syndrome occurance after acute COVID-19 disease in outpatients treated with and without cholecalciferol between 01/01/2020 and 31/12/2022
Analyse the rates of SARS-CoV-2 infection occurrence after anti-COVID-19 vaccination in patients treated with and without cholecalciferol. | to 01/01/2020 from 31/12/2022
  Analyse the rates of SARS-CoV-2 infection occurrence after anti-COVID-19 vaccination in oupatients treated with and without cholecalciferol between 01/01/2020 and 31/12/2022

CONTACTS AND LOCATIONS:
Locations (1):
- Luigi di Filippo, Milan, Italy